CLINICAL TRIAL: NCT01887730
Title: Can Intensified Hand Hygiene Decrease Morbidity and Lost Service Days in a Garrison
Brief Title: Hand Hygiene Intervention Study in Finnish Garrison
Acronym: VirusFight
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Organizational changes and lack of resources
Sponsor: Finnish Institute for Health and Welfare (Other Government)
Collaborators: Finnish Defense Forces (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: THL/81/6.05.00/2012
Record Dates: First submitted 2013-06-19; First posted 2013-06-27 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Infections
Keywords: Hand Hygiene; Communicable Diseases; Prevention
MeSH Terms: conditions — Infections; Communicable Diseases | interventions — Hand Disinfection; Soaps; Water; Ethanol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- arm 2 (Active Comparator): Hand washing with soap and water according to instructions. The effect of intervention is assessed by following occurrence of infections.
  Interventions: Behavioral: Hand washing with soap and water
- arm 0 (Placebo Comparator): No specific advice on hand hygiene. The effect of intervention is assessed by following occurrence of infections.
  Interventions: Behavioral: Control
- Arm 3 (Active Comparator): Hand cleaning with alcohol-containing hand rub
  Interventions: Behavioral: Hand cleaning with alcohol-containing hand rub

INTERVENTIONS:
Behavioral: Hand washing with soap and water — Can infections be prevented by hand washing with soap and water
  Arms: arm 2
Behavioral: Hand cleaning with alcohol-containing hand rub — Can infections be prevented by hand cleaning with alcohol-containing hand rub. Effect of intervention is assessed by following occurrence of infections
  Arms: Arm 3
Behavioral: Control
  Arms: arm 0

SUMMARY:
In this study the investigators aim to elucidate the possibility to reduce occurrence of infectious diseases in a garrison with enhanced and guided hand hygiene. The investigators will study occurrence and transmission of infections. In addition, the investigators will find out the causative agents of infections in a garrison with virological analyses of naso-pharyngeal and fecal specimens. The costs of lost service days and other expenses due to infectious diseases will be evaluated with a cost analysis study.

ELIGIBILITY:
Inclusion Criteria:

* willingness to attend to the study

Exclusion Criteria:

* skin diseases which prevent using hand disinfectants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1120 (Actual)
Dates: Start 2012-01; Primary Completion 2013-09 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Number of infection episodes during basic training period. The periods when a person has been in duty in spite of the infection will be included. | 8 weeks

SECONDARY OUTCOMES:
Length of distinct infection episodes due to infectious disease | 8 weeks
Length of distinct absence episodes due to infectious disease. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carita Savolainen-Kopra, Principal Investigator — Finnish Institute for Health and Welfare
Locations (1):
- Vekaranjärvi garrison, Kouvola, Finland